CLINICAL TRIAL: NCT07226726
Title: Mesenchymal Stem Cell Exosome Treatment of Congenital Myasthenic Syndrome
Brief Title: Patients With Congenital Myasthenic Syndrome Will be Treated With Mesenchymal Stem Cell Exosome Solution
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOREM2025-CMS1
Record Dates: First submitted 2025-11-05; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Congenital Myasthenic Syndrome
Keywords: exosomes; secretome; Congenital Myasthenic Syndrome
MeSH Terms: conditions — Myasthenic Syndromes, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental)
  Interventions: Biological: AlloEx exosomes

INTERVENTIONS:
Biological: AlloEx exosomes — This is an intranasal treatment of exosomes derived from mesenchymal stem cells.

SUMMARY:
Patients with Congenital Myasthenic Syndrome will be treated with Mesenchymal Stem Cell Exosome solution.

DETAILED DESCRIPTION:
Single Arm non-controlled study. Patients are prospectively evaluated then treated. Outcomes are tracked after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients will need a diagnosis of Congenital Myasthenic Syndrome by a licensed physician.
* Patients must be able to provide informed consent, or have a guardian who does.
* Patient must be able to travel to the site of treatment.

Exclusion Criteria:

* Patients will be excluded from the trial if they are pregnant or have active cancer (malignancy) at the screening consultation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen Saturation | From enrollment to 6 months after treatment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - Prodromos Stem Cell Institute, Naples, Florida
  - Prodromos Stem Cell Institute, Irving, Texas
- Medical Surgical Associates Center, St John's, Antigua and Barbuda